CLINICAL TRIAL: NCT05280210
Title: Patient-derived Tumor-like Cell Clusters (PTC) in Personalizing Neoadjuvant Therapy for Patients With Advanced Gastrointestinal Tumor: A Prospective, Open-label and Randomized Study
Brief Title: PTC in Personalizing Neoadjuvant Therapy for Patients With Advanced Gastrointestinal Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, Head of Beijing Cancer Hospital, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PKUCH-PTC
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Gastrointestinal Neoplasms
Keywords: neoadjuvant; chemotherapy
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant therapy based on PTC drug screening (Experimental): Patients will receive neoadjuvant therapy based on PTC drug screening. The regimen is complied with NCCN and CSCO guidelines. PD-1 inhibitor will be used if effective in drug screening.
  Interventions: Other: PTC drug screening
- Neoadjuvant therapy based on clinical experience (No Intervention): Patients will receive neoadjuvant therapy based on clinical experience. The regimen is complied with NCCN and CSCO guidelines.

INTERVENTIONS:
Other: PTC drug screening — PTC is an in vitro tumor model, which serves as a structural and functional unit recapitulating the original tumors in genotype, phenotype, and drug response. PTC will be used in drug screening.
  Arms: Neoadjuvant therapy based on PTC drug screening

SUMMARY:
To explore the value of PTC drug screening technique in selecting neoadjuvant therapy for advanced gastrointestinal cancer.

DETAILED DESCRIPTION:
In this study, patients diagnosed with advanced gastrointestinal cancer including locally advanced gastric cancer, locally advanced colorectal cancer and colorectal cancer with liver metastasis. Tumor sample will be collected by endoscopy biopsy, needle biopsy or surgery, which will used for PTC drug screening.

Patients will be randomized to two groups. Patients in experiment group will receive neoadjuvant therapy based on PTC drug screening, and patients in control group will receive neoadjuvant therapy based on clinical experience. 2-4 cycles of neoadjuvant therapy will be administered. Patients appropriate for surgery will receive radical surgery after neoadjuvant therapy. Pathological response will be compared primarily between these two groups.

This is a randomized controlled, open-label and sequential designed clinical trial. All neoadjuvant therapy used in this study or for PTC drug screening comply with NCCN (National comprehensive cancer network) or CSCO (Chinese Society of Clinical Oncology) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed of gastrointestinal adenocarcinoma by biopsy
* existence of initially resectable lesions evaluated by investigators
* indications of neoadjuvant chemotherapy including: 1) locally advanced gastric cancer cT1-2N1-3M0 & cT3-4N0-3M0; 2) locally advanced colorectal cancer cT3-4 or N+; 3)colorectal carcinoma with synchronous liver metastases: CRS≤2; 4)other patients who are considered to be appropriate to receive neoadjuvant chemotherapy determined by MDT
* never receive any tumor related treatment including chemotherapy, radiotherapy, and immune therapy
* never diagnosed of other malignancies
* able to tolerate chemotherapy
* ECOG≤2
* life expectance >6 months
* at least 1 measurable lesions(according to RECIST 1.1)
* informed consent

Exclusion Criteria:

* pregnant or lactating women
* participating in other clinical trials within 6 months
* MSI-H or dMMR or EBER(+)
* lesion located within 10cm from anal margin
* severe liver dysfunction
* severe renal dysfunction
* cognitive disorder, mental disease or poor compliance
* allergic to known chemotherapeutic agents
* other conditions not suitable to participate in this trial determined by investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate(pCR) | immediately evaluated after surgery
  having no invasive cancer left in the resected sample

SECONDARY OUTCOMES:
pathological response rate | immediately evaluated after surgery
  tumor regression grade 0-2
objective response rate(ORR) | evaluated by imaging before surgery
  CR+PR according to RECIST 1.1
disease control rate(DCR) | evaluated by imaging before surgery
  CR+PR+SD according to RECIST 1.1
R0 resection rate | immediately evaluated after surgery
  microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed
prediction accuracy of PTC | immediately evaluated after surgery
  consistency between the effect of neoadjuvant chemotherapy and the result of PTC assay

CONTACTS AND LOCATIONS:
Overall Officials: Aiwen Wu, M.D., Study Director — Peking University Cancer Hospital & Institute